CLINICAL TRIAL: NCT01565174
Title: The Pharmaco-genetic and Brain Mechanisms Associated With Cannabis- Induced Psychosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, VEINSHTEIN AVIV, Senior Research Fellow, Hadassah Medical Organization
Other Study IDs: 0541-11-HMO-CTIL
Record Dates: First submitted 2012-03-26; First posted 2012-03-28 (Estimated); Last update posted 2012-04-03 (Estimated); Status verified 2012-04

CONDITIONS: Cannabis Dependence; Psychosis
Keywords: cannabis; THC; COMT; psychosis; D2
MeSH Terms: conditions — Marijuana Abuse; Psychotic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Samples of DNA will be taken from saliva of participants
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- High activity COMT: Carriers of high activity COMT158Val allele who are expected to show higher THC-induced meso-limbic DA release
- Low activity COMT: Carriers of low activity COMT 158Met homozygotes are expected to release low amount of dopamine after smoking a cigarette with THC

SUMMARY:
There is growing evidence of high rates of substance use disorders among individuals with psychotic disorders especially in young people with predisposition for psychosis. There is some genetic evidence that carriers of the valine158 allele of the catechol-O-methyltransferase (COMT) gene had increased risk to exhibit psychotic symptoms and to develop schizophrenia if they used cannabis by the age of 18. It was also shown that carriers of the COMT val/val genotype were most sensitive to THC-induced psychotic experiences but this was conditional on pre-existing susceptibility to psychosis. The investigators propose to use brain-imaging and molecular genetics to investigate whether genetic factors may contribute to the THC-induced dopamine release and possibly to cannabis- induced psychosis.

DETAILED DESCRIPTION:
Genetic association study will be performed in 100 young cannabis users (age 18-26 years) for genes that are related to the neurotransmitters dopamine (D2, DAT, COMT), GABA, glutamate and the cannabinoid receptor CB1. Out of this cohort, 24 male subjects without history of cannabis or drug-induced psychosis will undergo brain imaging procedure in order to measure THC-induced dopamine release using [11C] Raclopride in PET imaging. Carriers of high activity COMT158Val allele are expected to show higher meso-limbic DA release than carriers of low activity COMT 158Met homozygotes and after smoking a cigarette with THC which in turn are thought to underlie the risk for THC-induced psychotic symptoms. The aim of the present study is to evaluate the relationship between the COMT genotype and cannabis-induced meso-limbic dopamine release as measured by D2 occupancy. In addition, the association between predisposition to psychosis, age of onset of cannabis dependence, and genotype of COMT and other neurotransmitters-related genes will be evaluated. Such finding could provide novel pharmaco-genetic explanation for the psychogenic effects of cannabis in vulnerable individuals.

ELIGIBILITY:
Inclusion Criteria:

* age 18-26 meeting DSM-IV-TR (American Psychiatric Association, 1994) diagnosis of THC dependence will be recruited from the general population by advertisement in the newspapers.

Exclusion Criteria:

* dependence on other substances or alcoholism
* a history of CNS disease
* a history of infection that might affect CNS (HIV, syphilis, cytomegalovirus, herpes)
* a history of head injury with loss of consciousness and pregnancy

Ages: 18 Years to 26 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: 100 current users of cannabis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Genetic variations of Dopamine, GABA, glutamate, cannabis CB1 receptor | 2 years
  DNA will be extracted from saliva of participants. Genetic variations of DA, GABA, glutamate and cannabis receptor CB1 will be coded.

SECONDARY OUTCOMES:
Measures of dopamine D2 receptor occupancy before and after smoking a cigarette containing THC. | 2 years
  Participants will be studied in a brain imaging study using [C 11] raclopride radioligand in Positron Emission Tomography (PET). Measures of D2 receptor occupancy will be taken at baseline and after smoking a cigarette containing 15 mg THC.

CONTACTS AND LOCATIONS:
Overall Officials: Aviv Weinstein, Ph.D, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel, Jerusalem, Israel